CLINICAL TRIAL: NCT04490798
Title: A Retrospective Longitudinal Cohort Study to Determine the Effectiveness of Integrated a Clinical Pathway Approach for Chronic Pain Treatment With Acupuncture in a Pain Clinic
Brief Title: Effectiveness of Acupuncture Clinical Pathway
Acronym: ACUPATHWAY
Status: Completed | Type: Observational
Sponsor: Hospital Son Llatzer (Other)
Responsible Party: Principal Investigator, Javier Mata, Principal Investigator, Hospital Son Llatzer
Other Study IDs: ACUPATHWAY.R.1
Record Dates: First submitted 2020-07-26; First posted 2020-07-29 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Chronic Pain; Lumbar Back Pain; Osteoarthritis, Knee; Headache; Shoulder Pain; Cervicalgia; Musculoskeletal Pain
Keywords: acupuncture treatment; clinical pathway
MeSH Terms: conditions — Chronic Pain; Low Back Pain; Osteoarthritis, Knee; Headache; Shoulder Pain; Neck Pain; Musculoskeletal Pain | interventions — Electroacupuncture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Lumbar back pain: Patients with lumbar back pain treated following the Acupuncture Treatment Clinic Pathway.
  Interventions: Procedure: Electroacupuncture
- Musculoskeletal pain: Patients with musculoskeletal pain treated following the Acupuncture Treatment Clinic Pathway.
  Interventions: Procedure: Electroacupuncture
- Cervicalgia: Patients with cervicalgia treated following the Acupuncture Treatment Clinic Pathway.
  Interventions: Procedure: Electroacupuncture
- Knee osteoarthritis: Patients with knee osteoarthritis treated following the Acupuncture Treatment Clinic Pathway.
  Interventions: Procedure: Electroacupuncture
- Headache: Patients with headache treated following the Acupuncture Treatment Clinic Pathway.
  Interventions: Procedure: Electroacupuncture
- Shoulder pain: Patients with shoulder pain treated following the Acupuncture Treatment Clinic Pathway.
  Interventions: Procedure: Electroacupuncture

INTERVENTIONS:
Procedure: Electroacupuncture — The electro-acupuncture device was a biphasic pulse generator. It was used with maximum tolerable intensity of current and a frequency of 3 Hz. The points were selected according to the Traditional Chinese Medicine meridian theory to treat the different painful syndromes. Just as in a regular acupuncture treatment, needles are inserted into acupuncture points but small crocodile clips are then attached to the ends of needles to connect them to an electro-acupuncture device. In traditional acupuncture the inserted needles are manually vibrated to induce a response whilst in electro-acupuncture the bi-phasic current results in a constant (controlled) vibration of the needles and a direct electrical stimulation.

SUMMARY:
The study will be described the development and implementation of the Clinical pathway (CPW) for acupuncture treatment in the management of patients with some chronic pain conditions. The effectiveness of this CPW will be explored in this study through retrospective analysis of clinical outcomes after administration of acupuncture treatment summarised in the guidelines.

DETAILED DESCRIPTION:
This longitudinal, observational, retrospective study included adults (>18 years) with common chronic pain condition treated at the Son Llàtzer University Hospital Pain Clinic, in Palma de Mallorca, Spain, from January 2015 to December 2018. All patients received treatment according to the Acupuncture Clinical Pathway developed. The primary outcome measures will be a change in pain intensity measured by VAS for pain at the completion of treatment. Number of responder patients, reduction of pain medication intake, improve of quality of live scale, sleep quality index and scale of anxiety and depression after treatment are also to be included in the study.

The purpose of this study is to assess the effectiveness of integrated a clinical pathway approach for chronic pain treatment with acupuncture in a Pain Clinic.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (>18 years) Acupuncture treatment for chronic pain (cervicalgia, low back pain, knee osteoarthritis, shoulder pain, headache or musculoskeletal pain), Applying Acupuncture treatment Clinical Pathway and completed at least 50% of the medical appointments.

Exclusion Criteria:

Inclusion Criteria:

Adult patients (>18 years) Acupuncture treatment for chronic pain (cervicalgia, low back pain, knee osteoarthritis, shoulder pain, headache or musculoskeletal pain), Without applying Acupuncture treatment Clinical Pathway or not completed at least 50% of the medical appointments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>18 years), who received acupuncture treatment for chronic pain (cervicalgia, low back pain, knee osteoarthritis, shoulder pain, headache or musculoskeletal pain), applying Acupuncture Treatment Clinical Pathway.
Sampling Method: Probability Sample
Enrollment: 3245 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity measured by VAS for pain at the completion of treatment | Baseline and after the completion of treatment at 4 months
  Overall average pain intensity over the last month will be assessed by a continuous scale comprised of a horizontal line, anchored by 'no pain' (score of 0) and 'worst imaginable pain' (score of 100 (100 mm scale)

SECONDARY OUTCOMES:
Number of responder patients to the acupuncture treatment. | Baseline, 1 month and after the completion of treatment at 4 months
  Responders will be defined as patients with a reduction of pain scores of more than 30%, decreasing medication intake or improving quality of live scale (≥ 20%), sleep quality index (≥ 30%) following our Clinical Pathway.
Reduction of pain medication intake after treatment | Baseline, 1 month and after the completion of treatment at 4 months
  Analgesic medicine use will be obtained with a questionnaire elaborated according to the European Health Interview Survey (EUROHIS) recommendations. Subjects will be asked (1) about the prescription medicine their general practitioner may have prescribed for them ('Have you taken any pain medicine prescribed by your general practitioner?') as well as any medication not prescribed by their general practitioner ('Have you taken any pain medicine not prescribed by your general practitioner') and (2) whether their prescribed and non-prescribed pain medication use has increased or decreased.
Improve of quality of live scale after treatment | Baseline, 1 month and after the completion of treatment at 4 months
  Patient-related quality of live by SF-12 measured. The Spanish version validated by Schmidt S et al is used
Improve sleep quality index after treatment | Baseline, 1 month and after the completion of treatment at 4 months
  Measured with the Pittsburgh Sleep Quality Index (PSQ). The Spanish version validated by Hita-Contreras F et al is used
Improve of scale of anxiety and depression after treatment | Baseline, 1 month and after the completion of treatment at 4 months
  Levels of depression and anxiety will be measured with the Goldberg Anxiety and Depression Scale. The Spanish version validated by Montón et al is used.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Mata, MD, Principal Investigator — Anaesthesia Department, Son Llàtzer University Hospital. Palma, Spain
Locations (1):
- Son Llatzer University Hospital, Palma, Balear Islands, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eisenberg DM, Davis RB, Ettner SL, Appel S, Wilkey S, Van Rompay M, Kessler RC. Trends in alternative medicine use in the United States, 1990-1997: results of a follow-up national survey. JAMA. 1998 Nov 11;280(18):1569-75. doi: 10.1001/jama.280.18.1569. PMID 9820257
- [Background] Vickers AJ, Cronin AM, Maschino AC, Lewith G, MacPherson H, Foster NE, Sherman KJ, Witt CM, Linde K; Acupuncture Trialists' Collaboration. Acupuncture for chronic pain: individual patient data meta-analysis. Arch Intern Med. 2012 Oct 22;172(19):1444-53. doi: 10.1001/archinternmed.2012.3654. PMID 22965186
- [Background] Lee MS, Ernst E. Acupuncture for pain: an overview of Cochrane reviews. Chin J Integr Med. 2011 Mar;17(3):187-9. doi: 10.1007/s11655-011-0665-7. Epub 2011 Feb 27. PMID 21359919
- [Background] Vickers AJ, Linde K. Acupuncture for chronic pain. JAMA. 2014 Mar 5;311(9):955-6. doi: 10.1001/jama.2013.285478. PMID 24595780
- [Background] Dowell D, Haegerich TM, Chou R. CDC Guideline for Prescribing Opioids for Chronic Pain--United States, 2016. JAMA. 2016 Apr 19;315(15):1624-45. doi: 10.1001/jama.2016.1464. PMID 26977696
- [Background] Qaseem A, Wilt TJ, McLean RM, Forciea MA; Clinical Guidelines Committee of the American College of Physicians; Denberg TD, Barry MJ, Boyd C, Chow RD, Fitterman N, Harris RP, Humphrey LL, Vijan S. Noninvasive Treatments for Acute, Subacute, and Chronic Low Back Pain: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2017 Apr 4;166(7):514-530. doi: 10.7326/M16-2367. Epub 2017 Feb 14. PMID 28192789
- [Background] Camm AJ, Fox KAA. Strengths and weaknesses of 'real-world' studies involving non-vitamin K antagonist oral anticoagulants. Open Heart. 2018 Apr 21;5(1):e000788. doi: 10.1136/openhrt-2018-000788. eCollection 2018. PMID 29713485
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) Statement: guidelines for reporting observational studies. Int J Surg. 2014 Dec;12(12):1495-9. doi: 10.1016/j.ijsu.2014.07.013. Epub 2014 Jul 18. PMID 25046131
- [Background] Nosikov A , Gudex C . eds. EUROHIS:, "Developing common instruments for health surveys. Amsterdam: IOS Press, 2003.".
- [Background] Monton C, Perez Echeverria MJ, Campos R, Garcia Campayo J, Lobo A. [Anxiety scales and Goldberg's depression: an efficient interview guide for the detection of psychologic distress]. Aten Primaria. 1993 Oct 15;12(6):345-9. Spanish. PMID 8218816
- [Background] Schmidt S, Vilagut G, Garin O, Cunillera O, Tresserras R, Brugulat P, Mompart A, Medina A, Ferrer M, Alonso J. [Reference guidelines for the 12-Item Short-Form Health Survey version 2 based on the Catalan general population]. Med Clin (Barc). 2012 Dec 8;139(14):613-25. doi: 10.1016/j.medcli.2011.10.024. Epub 2012 Jan 11. Spanish. PMID 22244683
- [Background] Hita-Contreras F, Martinez-Lopez E, Latorre-Roman PA, Garrido F, Santos MA, Martinez-Amat A. Reliability and validity of the Spanish version of the Pittsburgh Sleep Quality Index (PSQI) in patients with fibromyalgia. Rheumatol Int. 2014 Jul;34(7):929-36. doi: 10.1007/s00296-014-2960-z. Epub 2014 Feb 8. PMID 24509897
- [Background] Dworkin RH, Turk DC, McDermott MP, Peirce-Sandner S, Burke LB, Cowan P, Farrar JT, Hertz S, Raja SN, Rappaport BA, Rauschkolb C, Sampaio C. Interpreting the clinical importance of group differences in chronic pain clinical trials: IMMPACT recommendations. Pain. 2009 Dec;146(3):238-244. doi: 10.1016/j.pain.2009.08.019. PMID 19836888
- [Background] Vickers AJ, Vertosick EA, Lewith G, MacPherson H, Foster NE, Sherman KJ, Irnich D, Witt CM, Linde K; Acupuncture Trialists' Collaboration. Acupuncture for Chronic Pain: Update of an Individual Patient Data Meta-Analysis. J Pain. 2018 May;19(5):455-474. doi: 10.1016/j.jpain.2017.11.005. Epub 2017 Dec 2. PMID 29198932
- [Background] Herman JP, Figueiredo H, Mueller NK, Ulrich-Lai Y, Ostrander MM, Choi DC, Cullinan WE. Central mechanisms of stress integration: hierarchical circuitry controlling hypothalamo-pituitary-adrenocortical responsiveness. Front Neuroendocrinol. 2003 Jul;24(3):151-80. doi: 10.1016/j.yfrne.2003.07.001. PMID 14596810
- [Background] Harris RE, Zubieta JK, Scott DJ, Napadow V, Gracely RH, Clauw DJ. Traditional Chinese acupuncture and placebo (sham) acupuncture are differentiated by their effects on mu-opioid receptors (MORs). Neuroimage. 2009 Sep;47(3):1077-85. doi: 10.1016/j.neuroimage.2009.05.083. Epub 2009 Jun 6. PMID 19501658
- [Background] Zubieta JK, Stohler CS. Neurobiological mechanisms of placebo responses. Ann N Y Acad Sci. 2009 Mar;1156:198-210. doi: 10.1111/j.1749-6632.2009.04424.x. PMID 19338509
- [Background] Lee SC, Yin SJ, Lee ML, Tsai WJ, Sim CB. Effects of acupuncture on serum cortisol level and dopamine beta-hydroxylase activity in normal Chinese. Am J Chin Med. 1982;10(1-4):62-9. doi: 10.1142/S0192415X82000117. PMID 7183209
- [Background] Schneider A, Weiland C, Enck P, Joos S, Streitberger K, Maser-Gluth C, Zipfel S, Bagheri S, Herzog W, Friederich HC. Neuroendocrinological effects of acupuncture treatment in patients with irritable bowel syndrome. Complement Ther Med. 2007 Dec;15(4):255-63. doi: 10.1016/j.ctim.2006.12.002. Epub 2007 Feb 20. PMID 18054727
- [Background] Tsigos C, Chrousos GP. Hypothalamic-pituitary-adrenal axis, neuroendocrine factors and stress. J Psychosom Res. 2002 Oct;53(4):865-71. doi: 10.1016/s0022-3999(02)00429-4. PMID 12377295
- [Background] Lawal AK, Rotter T, Kinsman L, Machotta A, Ronellenfitsch U, Scott SD, Goodridge D, Plishka C, Groot G. What is a clinical pathway? Refinement of an operational definition to identify clinical pathway studies for a Cochrane systematic review. BMC Med. 2016 Feb 23;14:35. doi: 10.1186/s12916-016-0580-z. PMID 26904977
- See also: Wide-ranging online data for epidemiologic research (WONDER). , "Atlanta, GA: CDC, National Center for Health Statistics," 2016. [Online]. Available: http://wonder.cdc.gov.. [Accessed 7 july 2020]. — https://wonder.cdc.gov